CLINICAL TRIAL: NCT03183024
Title: Treatment of Chronic Urticarial Unresponsive to H1-antihistamines With an Anti-IL5Ralpha Monocloncal Antibody
Brief Title: Treatment of Chronic Urticarial Unresponsive to H1-antihistamines With an Anti-IL5Ralpha Monoclonal Antibody
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jonathan A. Bernstein, MD (Other)
Responsible Party: Sponsor-Investigator, Jonathan A. Bernstein, MD, PI/ co-owner, Bernstein Clinical Research Center
Organization: Bernstein Clinical Research Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAIRB-17-0036
Record Dates: First submitted 2017-05-25; First posted 2017-06-09 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): placebo for benralizumab sc given during run-in phase
  Interventions: Biological: placebo
- benralizumab (Experimental): benralizumab sc once a month for 3 months for subjects who meet inclusion/exclusion criteria after run-in phase
  Interventions: Biological: benralizumab

INTERVENTIONS:
Biological: benralizumab — open-label treatment
  Arms: benralizumab
Biological: placebo — sterile water to mimic benralizumab
  Arms: placebo

SUMMARY:
Study to determine the efficacy of benralizumab when compared to placebo in patients with chronic hives that do not respond to antihistamine treatment

DETAILED DESCRIPTION:
Subjects with chronic hives that do not respond to antihistamine treatment and have hives of unknown cause will be eligible. Subjects who meet the inclusion/exclusion criteria after the run-in phase will receive 3 doses of study medication. The study also involved blood draws and a punch biopsy of a hive

ELIGIBILITY:
Inclusion Criteria:

* hives for over 6 weeks of unknown cause hives most days of the despite use of antihistamines

Exclusion Criteria:

* hives due to known reasons history of cancer pregnant or nursing History of HIV or Hepatitis recent parasitic infection currently or have received treatment with a monoclonal antibody

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
change in urticarial activity score averaged over 7 days- no units | through study completion, up to 7 months
  subject completed form

SECONDARY OUTCOMES:
change in blood anti-FCER1 level (kU/l) | through study completion, up to 7 months
  specific lab test
change in blood anti-TPO level (IU/L) | through study completion, up to 7 months
  specific blood test
change in Blood ECP level (ug/L) | through study completion, up to 7 months
  specific blood test
change in blood eotaxin level (pg/ml) | through study completion, up to 7 months
  specific blood test
change in RNA testing | through study completion, up to 7 months
  gene expression profile using RNA-sequencing in skin biopsy samples (lesional vs non-lesional skin) (log 2 fold-change)
change in skin biopsy inflammatory cell counts | through study completion, up to 7 months
  inflammatory cell count in skin biopsy (number of cells/sq mm)
change in cytokine quantification in skin biopsy (units/mL) | through study completion, up to 7 months
  skin biopsy

OTHER OUTCOMES:
adverse events | through study completion, up to 7 months
  adverse events
change in blood pressure | through study completion, up to 7 months
  blood pressure- mm Hg
change in pulse rate | through study completion, up to 7 months
  pulse rate- bpm
change in blood urea nitrogen | through study completion, up to 7 months
  blood urea nitrogen lab test - mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Bernstein Clinical Research Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided